CLINICAL TRIAL: NCT05977686
Title: Point-of-Care Hemoglobin Testing in Pregnant Patients
Brief Title: Hemoglobin Testing in Pregnant Patients
Acronym: Prosp Anemia
Status: Recruiting | Type: Observational
Sponsor: George Washington University (Other)
Collaborators: Inova Health Care Services (Other)
Responsible Party: Principal Investigator, Homa K. Ahmadzia, PI, Inova Health Care Services
Other Study IDs: NCR234874
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Post Partum Hemorrhage; Anemia of Pregnancy
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Masimo Root Radical 7 Pulse CO-Oximeter — The Masimo device is non-invasive and placed externally on a patient's finger to generate an estimation of a patient's hemoglobin value.
Device: HemoCue Hb 801 — The HemoCue® device is a minimally-invasive device that relies on the finger prick method to get a capillary hemoglobin measurement.

SUMMARY:
The project is a prospective observational study aimed to assess and to validate the use of point-of-care hemoglobin testing in pregnancy. Point-of-care hemoglobin testing has the potential to (1) increase access to hemoglobin monitoring in pregnancy in low resource settings, (2) increase availability of hemoglobin monitoring in anemic patients, and (3) provide immediate results for real-time patient counseling and intervention. However, to date, point-of-care hemoglobin testing devices have not yet been studied for use in an ambulatory obstetric population. The Masimo device is a Root Radical 7 Pulse CO-Oximeter, manufactured by Masimo, Inc. This device is non-invasive and placed externally on a patient's finger to generate an estimation of a patient's hemoglobin value. The HemoCue® device is a minimally-invasive device that relies on the finger prick method to get a capillary hemoglobin measurement, and The Rubby is a mobile application based platform that uses a photo of the participants nailbed to estimate hemoglobin values. Participants in this study will be approached at the Obstetrics and Gynecology clinics at George Washington Medical Faculty Associates. Point-of-care hemoglobin measurements will be assessed using the non-invasive Masimo device along with minimally-invasive hemoglobin HemoCue® Hb 801 device and compared to traditional venipuncture hemoglobin testing.

DETAILED DESCRIPTION:
This will be a prospective, observational study for which aim to recruit 200 patients over the study period. Patients will be approached at one of the MFA Obstetrics and Gynecology clinics. Once consented, they will be approached at least two time-points during their antenatal care as below:

1. OB new/ first prenatal visit (usually between 12-18 weeks of gestation)
2. OB return visit (usually between 24-28 weeks of gestation)

May need to get more Hb time-points readings (up to five readings) if the patient will be diagnosed with anemia at any of the previously mentioned visits or will be scheduled to have more blood draws during the prenatal care period. At each time-point visit, we plan to talk with the provider of the patient about the study. Then the study protocol and the recruitment process with the patient will be discussed. If the patient consents, the researchers will coordinate with the lab personnel the exact time of the routinely ordered blood draw (as a part of the subject's antenatal care) to determine the appropriate time to get the Hb readings using the devices (preferrably, right before the venipuncture). To obtain the readings, a study research coordinator will apply a disposable probe (Rainbow R1 25 adult adhesive sensor) connected to a Radical-7 co-oximeter sensor on the ring finger of the same arm of the venipuncture, shielded by an opaque covering to eliminate intereference from ambient light to obtain the SpHb reading. In addition, during in the same setting, we will ask for a finger prick capillary sample to get the Hemocue Hb reading as well (the same side will be used). Both readings will be tabulated in a case report form and the standard lab hemoglobin reading will be added to them once received. This is how it will validate the performance of the Masimo and the Hemocue devices with the routine lab test results. Additionally, the researchers will collect demographics, procedure-specific and some antenatal-care variables including vitals, gestational age and the exact date and time of the records at each time point visit, using a well-structured case report form.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ages 18-50 years old

Exclusion Criteria:

* Patients with hemoglobinopathies (qualitative defects, sickle-cell anemia) and hemoglobin synthesis disorders (quantitative defects such as thalassemia)
* Patients with peripheral vascular diseases and skin conditions that affect blood vessels in the digit
* Patients with hyperbilirubinemia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women ages 18-50 years old
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the devices in all obstetric patients | 2024
Ability of point-of-care hemoglobin testing devices to detect anemia (Hemoglobin less than 11 mg/dL) or severe anemia (Hemoglobin less than 9 mg/dL). | 2024
Subgroup analysis: by gestational age categories presence or absence of anemia as defined by the gold standard venipuncture | 2024
Patient perception of testing methods | 2024

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - George Washington University, Washington D.C., District of Columbia
  - Inova Health System, Falls Church, Virginia